CLINICAL TRIAL: NCT01697930
Title: A Phase I Study: PET Imaging of Cancer Patients Using [18F] 4-L-Fluoroglutamine (2S,4R)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-168
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Solid Malignancy; Lymphoma
Keywords: PET Imaging; 18F] 4-L-Fluoroglutam (2S,4R); 12-168
MeSH Terms: conditions — Lymphoma

ARMS (1):
- [18F] 4-L-Fluoroglutamine (2S,4R) (Experimental): This pilot, first in-human microdose PET trial of the positron-emitting agent [18F] 4-L-Fluoroglutamine (2S,4R) will be an open-label study. The [18F] 4-L-Fluoroglutamine (2S,4R) agent will be administered by bolus intravenous injection. In all study patients, the pharmacokinetics, metabolism, and biodistribution of [18F] 4-L-Fluoroglutamine (2S,4R) will be evaluated by non-invasive blood- and PET-based assays, at multiple time points (see Table 1,) during one day. Eligible patients optionally can participate in the study twice, on a separate date, receiving a second radiotracer microdose of [18F] 4-L-Fluoroglutamine (2S,4R), followed by non-invasive blood- and PET-based assays. At the discretion of the investigator, scan 3 can be waived.
  Interventions: Drug: [18F] 4-L-Fluoroglutamine (2S,4R)

INTERVENTIONS:
Drug: [18F] 4-L-Fluoroglutamine (2S,4R) — Thirty cancer patients will receive an injection of a 0.5 to 7.5mCi of [18F] 4-LFluoroglutamine (2S,4R) , followed by serial PET/CT scanning and blood draws, (at the direction of the investigator) over a period of 3.5 hours, on a single day. Each patient will be offered the opportunity to repeat the [18F] 4-L-Fluoroglutamine (2S,4R) injection and subsequent set of post-injection PET-CT scans, once, on a separate date. At the discretion of the investigator, scan 3 can be waived. Immediately prior to injection of the radiotracer, a blood sample will be obtained for measurement of serum glutamine level. The serum glutamine level will be assayed, if necessary, as part of an amino acid screen assay.

SUMMARY:
This is a Phase I study. This study is the first time that a new experimental drug called 18FFluoroglutamine, or F-Glutamine, is being used in people. F-Glutamine is a drug designed to be used with PET scanners that can 'see' where F-Glutamine goes in the body, after its injected. PET scanners are one of the kinds of scanners you normally find in a hospital radiology department. The researchers have found that tumors in animals absorb F-Glutamine. The researchers believe that scans with F-Glutamine might be able to find tumors in patients.

This first in-human study is being done to see how long F-Glutamine lasts in the blood, when it is given to people in tiny amounts by an injection, and to see where F-Glutamine goes in the body. If the results of this trial are good, then the study doctors plan to use F-Glutamine in another trial to see if scans with F-Glutamine are better for finding tumors compared to the standard types of scans that doctors use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of histologically-confirmed solid malignancy and/or lymphoma (histology confirmed by MSKCC Department of Pathology.) Disease measurable or evaluable as defined by RECIST 1.1 or other tumor response criteria from an MSKCC IRB-approved clinical research protocol. NOTE: Study patients do not need to be participating in an MSKCC approved clinical trial prior to study recruitment.
* Age between 21-90
* Negative serum pregnancy test for female patients of childbearing age and potential (as defined by MSKCC Standards & Guidelines), from assays obtained <2 weeks prior to study enrollment. Patients will be advised against having unprotected sexual intercourse from the time of the negative serum pregnancy test until after completing their participation in the study.

Exclusion Criteria:

* Inability or refusal to have at least one peripheral intravenous line for intravenous access (as applicable to the day of [18F] 4-L-Fluoroglutamine (2S,4R) injection and blood draws.)
* Breast-feeding
* Refusal or inability to tolerate the scanning procedure (e.g., due to claustrophobia)
* Hepatic: from assays obtained <2 weeks prior to study enrollment For each patient, the upper limit of normal (ULN) value for a particular assay will be defined by the normal reference values of the laboratory that performed the assay.
* Bilirubin > 1.5 x (ULN)
* AST/ALT >2.5 x ULN
* Albumin < 3 g/dl
* GGT > 2.5 x ULN IF Alkaline phosphatase > 2.5 x ULN.
* Renal: Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min, from assays obtained <2 weeks prior to study enrollment
* Acute major illness (e.g., unstable cardiovascular condition, etc.)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetic profiles | 2 years
  The trial-design follows standard guidelines on collecting pharmacokinetic (PK) data for investigational radioactive drugs.1, 29-36 Animal [18F] 4-L-of [18F] 4-L-Fluoroglutamine (2S,4R). Fluoroglutamine (2S,4R) PK data provided a basis for the trial design. Sampling time-points were chosen (1) by anticipated exponential PK; with (2) allometry-based interspecies extrapolation of time-scales.37 As data is available from the first patients, suitability of the time-points will be re-examined. Blood samples will be centrifuged and the plasma pipetted, weighed and counted to determine the plasma time activity concentration curves (% injected dose/liter), as well as for metabolite analysis of the [18F] 4-L-Fluoroglutamine (2S,4R) compound (by radio-HPLC or other fit-for-purpose methodology).

SECONDARY OUTCOMES:
metabolism | 2 years
  Blood samples will be centrifuged and the plasma pipetted, weighed and counted to determine the plasma time activity concentration curves (% injected dose/liter), as well as for metabolite analysis of the [18F] 4-L-Fluoroglutamine (2S,4R) compound (by radio-HPLC or other fit-for-purpose methodology).
bio distribution | 2 years
  These data will be obtained in the form of serial PET imaging to detect and quantify changes [18F] 4-L-Fluoroglutamine (2S,4R) biodistribution at multiple time-points, as well as serial venous blood-assays. Our PET scans are routinely corrected for attenuation and scatter and adjusted for system sensitivity and provide quantitative images of the tracer concentration within the imaging field of view, which is often reported in terms of standardized uptake values (SUV) (= μCi found/gm tissue / μCi injected/gm body mass).
radiation dosimetry | 2 years
  OLINDA 1.1 software, an FDA-approved radiation-dosimetry software package42, 43 will be used to obtain absorbed dose & effective dose measurements. In brief, this entails its automated application of the MIRD formalism to the experimental time-integrated activity coefficients, with dose-factor values defined by standard isotope data and a hermaphroditic anthropomorphic model.34, 36, 38, 44 . OLINDA implements conventional biokinetic models of the urinary bladder and gastrointestinal tract to account for the dosimetric contribution of radioactive excreta.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dunphy, D.O., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Dunphy MPS, Harding JJ, Venneti S, Zhang H, Burnazi EM, Bromberg J, Omuro AM, Hsieh JJ, Mellinghoff IK, Staton K, Pressl C, Beattie BJ, Zanzonico PB, Gerecitano JF, Kelsen DP, Weber W, Lyashchenko SK, Kung HF, Lewis JS. In Vivo PET Assay of Tumor Glutamine Flux and Metabolism: In-Human Trial of 18F-(2S,4R)-4-Fluoroglutamine. Radiology. 2018 May;287(2):667-675. doi: 10.1148/radiol.2017162610. Epub 2018 Jan 31. PMID 29388903
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/